CLINICAL TRIAL: NCT02374255
Title: Improving Advanced Cancer Patient-Centered Care by Enabling Goals of Care Discussions
Brief Title: Improving Goals of Care Discussion in Advanced Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO 14-0082
Record Dates: First submitted 2015-02-09; First posted 2015-02-27 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Primary Stage IV Hepatobiliary; Esophageal; Colorectal Cancer; Glioblastoma; Cancer of Stomach; Cancer of Pancreas; Melanoma; Head or Neck Cancer; Stage III; Stage IV; Lung Cancers; Pancreatic Cancers
Keywords: Advanced cancer; goals of care; quality of care; end of life discussions
MeSH Terms: conditions — Colorectal Neoplasms; Glioblastoma; Stomach Neoplasms; Pancreatic Neoplasms; Melanoma; Head and Neck Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GoC intervention (Experimental): Oncologists trained using OncoTalk to have Goals of Care discussions.
  Interventions: Behavioral: GoC intervention
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: GoC intervention — Training of oncologists using OncoTalk to conduct Goals of Care discussions and measure impact on patient satisfaction.
  Other Names: Goals of Care discussions
  Arms: GoC intervention

SUMMARY:
The goal of this study is to increase and improve Goals of Care discussions for advanced cancer patients by training medical oncologists to conduct these discussions. The investigators will evaluate the GoC discussion's effects on patient satisfaction, receipt of treatment in line with preferences, use of aggressive treatment, and oncologist communication skill.

DETAILED DESCRIPTION:
Among advanced cancer patients, discussions about prognosis, goals of care (GoC) and end-of-life preferences improve quality of life of patients and reduce rates of hospital and ICU admission. Yet, few patients know their chemotherapy treatments will not cure their disease despite nearly all wishing to receive information- good & bad. Currently, 37% of advanced cancer patients have GoC clarifying discussions and when they do, it is often in the last 2 months of life when symptoms are uncontrollable and oncologists have no other treatments to offer. These discussions do not usually happen with the patient's personal oncologist. Current efforts to teach oncologists such skills are impractical, requiring a lot of time away from their office practice and do not take into account job pressures.

The goal of this study is to increase and improve GoC discussions for advanced cancer patients by training medical oncologists to conduct these discussions and evaluate its effects on patient satisfaction, receipt of care in line with preferences, aggressive care utilization, and oncologist communication skill.

The investigators will recruit 280 patients of which half will come from intervention doctors and the other from the control doctors. The investigators will train randomly selected oncologists to conduct GoC discussion. Patients will be surveyed at baseline within days of their GOC visit and at 6 months. Oncologists will be audio-taped at baseline and after training is complete to assess practice and skill to conduct GoC discussions.

Primary outcomes include patient reported conduct of and satisfaction with GoC discussion. Secondary outcomes include oncologist communication skills, feasibility of performing GoC in the outpatient setting, receipt of care in line with preferences, use of hospice, chemotherapy or ICU in the last 30 days of life.

ELIGIBILITY:
Inclusion Criteria:

* Men or women who are at least 21 years of age who have been diagnosed within one month with a pathologically confirmed advanced cancer who have an average of <2 y life expectancy (primary stage IV hepatobiliary, esophageal, colorectal, glioblastoma, gastric, pancreatic, melanoma, head & neck, or stage III or IV lung or pancreatic cancers) and are being treated at one of the participating hospital sites and speak English or Spanish.
* Oncologists who treat at least 2 advanced cancer patients per month at a study participating hospital will be enrolled into the study.

Exclusion Criteria:

* Patients who have seen an oncologist after undergoing first line treatment imaging as this group has a higher likelihood of having received a goals of care discussion.
* Men or women who do not speak English or Spanish will be excluded.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Bickell, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (4):
- United States (4):
  - Smilow Cancer Hospital, Yale Cancer Center, Yale University, New Haven, Connecticut
  - Mount Sinai Beth Israel, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Kings County Hospital Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Oncologists were not considered enrolled into the study.
Groups:
- Patients - GoC Intervention: Patients given OncoTalk GoC intervention
  GoC intervention: Training of oncologists using OncoTalk to conduct Goals of Care discussions and measure impact on patient satisfaction.
- Patients - Usual Care: Prospective control group where no intervention was given.
- Oncologists - GoC Intervention: Oncologists trained using OncoTalk to have Goals of Care discussions.
- Oncologists - Usual Care: Oncologists not trained using OncoTalk to have Goals of Care discussions.
Period: Overall Study
Arm/Group | Patients - GoC Intervention | Patients - Usual Care | Oncologists - GoC Intervention | Oncologists - Usual Care
Started | 155 | 110 | 11 | 11
Completed | 153 | 110 | 11 | 11
Not Completed | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data was collected for patient participants only
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients - GoC Intervention | Patients - Usual Care | Oncologists - GoC Intervention | Oncologists - Usual Care | Total
Number analyzed (Participants) | 155 | 110 | 0 | 0 | 265
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (12.3) | 65 (11.3) |  |  | 64 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 44 |  |  | 108
  Male | 91 | 66 |  |  | 157
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 21 |  |  | 50
  Not Hispanic or Latino | 126 | 89 |  |  | 215
  Unknown or Not Reported | 0 | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  |  | 0
  Asian | 8 | 3 |  |  | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
  Black or African American | 50 | 29 |  |  | 79
  White | 71 | 65 |  |  | 136
  More than one race | 26 | 13 |  |  | 39
  Unknown or Not Reported | 0 | 0 |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Perceived Increased Goals of Care Discussions
Description: Number of patient's perceptions that goals of care discussions were increased occurred as measured by GoC qualitative patient survey.
Time Frame: up to 6 months
Population: Data from patient participants only. Data not collected from Oncologists
Measure: Count of Participants; unit: Participants
Groups:
- Oncologist - GoC Intervention: Oncologists trained using OncoTalk to have Goals of Care discussions.
Arm/Group | Patients - GoC Intervention | Patients - Usual Care | Oncologist - GoC Intervention | Oncologists - Usual Care
Number analyzed (Participants) | 153 | 110 | 0 | 0
Participants | 43 | 34 |  |

2. Primary Outcome: Number of Patients Perception of Improved Goals of Care Discussions
Description: Number of Patient's satisfaction with the discussion of improved goals of care as measured by GoC qualitative patient survey.
Time Frame: up to 6 months
Population: Data collected for patient participants only
Measure: Count of Participants; unit: Participants
Groups:
- Patients - GoC Intervention: Patients given OncoTalk GoC intervention.
  GoC intervention: Training of oncologists using OncoTalk to conduct Goals of Care discussions and measure impact on patient satisfaction.
Arm/Group | Patients - GoC Intervention | Patients - Usual Care | Oncologists - GoC Intervention | Oncologists - Usual Care
Number analyzed (Participants) | 153 | 110 | 0 | 0
Participants | 70 | 65 |  |

3. Secondary Outcome: Communication Skills Training
Description: Oncologist's communication skills are tested and rated between 1 and 7, with higher number indicating the oncologists were more comfortable in demonstrating communication skills while having the Goals of Care discussion with their patients.
Time Frame: up to 6 months
Population: Participants represented are the oncologist's. Data collected for the oncologists only.
Measure: Mean (Standard Deviation); unit: number of skills tested
Groups:
- Oncologists - GoC Intervention: Oncologists trained using OncoTalk to have Goals of Care discussions.
  GoC intervention: Training of oncologists using OncoTalk to conduct Goals of Care discussions and measure impact on patient satisfaction.
Arm/Group | Oncologists - GoC Intervention | Oncologists - Usual Care | Patients - GoC Intervention | Patients - Usual Care
Number analyzed (Participants) | 11 | 11 | 0 | 0
number of skills tested | 3.7 (1.96) | 2.2 (1.08) |  |

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored/assessed
Description: Adverse events were not monitored/assessed
Arm/Group | Patients - GoC Intervention | Patients - Usual Care | Oncologists - GoC Intervention | Oncologists - Usual Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/55/NCT02374255/Prot_000.pdf
  • Statistical Analysis Plan (2015-02-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT02374255/SAP_001.pdf